CLINICAL TRIAL: NCT03989258
Title: Implementation of a Model for Personalised Risk-Based Breast Cancer Prevention and Screening
Brief Title: Personalised Risk-based Breast Cancer Prevention and Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tartu University Hospital (Other)
Collaborators: University of Tartu (Other); North Estonia Medical Centre (Other)
Responsible Party: Principal Investigator, Peeter Padrik, Director of the Cancer Center, Tartu University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: estPerMed 1, Breast
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Screening; Genetic risk; Polygenic risk score
MeSH Terms: conditions — Breast Neoplasms; Genetic Risk Score

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): High monogenic breast cancer risk
  Interventions: Diagnostic Test: Mammography outside official screening
- Cohort 2 (Active Comparator): High polygenic breast cancer risk
  Interventions: Diagnostic Test: Mammography outside official screening
- Cohort StMG (No Intervention): Standard mammography screening in age 50-69

INTERVENTIONS:
Diagnostic Test: Mammography outside official screening — Radiologic study
  Arms: Cohort 1; Cohort 2

SUMMARY:
This is a cohort study, applied research and T3 translational genomics to estimate the impact of genetic risk for breast cancer detection in the screening program. The study group base consists of 28 389 female participants, currently in the age-group 22-79, in the Biobank of Estonian Genome Centre. The study is aimed to demonstrate the usability of personalised approach for adjusting and stratifying screening recommendations, based on predicted genetic risk estimates for breast cancer in the situation, where the genome data could be available from all women who have given informed consent for that. The project includes both the detection of moderate and high hereditary breast cancer risk carriers as well as high risk polygenic risk-score (consisting several single nucleotide polymorphisms) carriers among healthy individuals for application of personalised prevention and screening strategies.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* Available NGS (WGS or WES) data for detection of breast cancer moderate to high genetic risk variants in BRCA1, BRCA2, TP53, STK11, PTEN, CDH1, ATM, PALB2, CHEK2, NBN, NF1 genes;
* Available genetic (WGS, genotyping) data for PRS calculation, participants in age 40-74 will be further selected;

Cohort 2:

* Available genotyping data;
* No available NGS data for BRCA1, BRCA2, TP53, STK11, PTEN, CDH1, ATM, PALB2, CHEK2, NBN, NF1 genes;
* Participants in the age group 40-74 with available genetic data for PRS calculation;

Cohort StMG:

• Female participants in Estonian Biobank in the age group 50-69 participating at least once in the current Estonian population-based screening program during 2016-2020.

Exclusion Criteria:

Cohort 1: breast cancer in the medical history; Cohort 2: breast cancer in the medical history. Cohort StMG: none.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28389 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of women in the population with genetically higher risk for breast cancer | 3 years

SECONDARY OUTCOMES:
Number of screen-detected breast cancers in different risk groups | 3-years

CONTACTS AND LOCATIONS:
Locations (2):
- Estonia (2):
  - Tartu University Hospital, Tartu, Tartu
  - The North Estonia Medical Centre, Tallinn

IPD SHARING:
Plan to Share IPD: Undecided